CLINICAL TRIAL: NCT05816148
Title: Leisure Physical Activity and Barriers to Physical Activity Among Members and Users of APF France Handicap
Brief Title: Leisure Physical Activity and Barriers to Physical Activity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut de Sante Parasport Connecte Synergies (Other)
Collaborators: Association des Paralysees de France (APF) (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-003
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Disabled Persons
Keywords: Exercise; Cross sectional studies; Social inclusion
MeSH Terms: conditions — Motor Activity; Social Inclusion | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Disabled persons: Members or users of APF France handicap
  Interventions: Other: Questionnaire survey

INTERVENTIONS:
Other: Questionnaire survey — On leisure physical activity, barriers to physical activity and quality of life.

SUMMARY:
People with disabilities are less physically active than the general population. Currently, the level of leisure physical activity of people who are members or users of APF France handicap and their barriers to physical activity are unknown. The APF France handicap association is a national movement for the defense and representation of people with disabilities and their families. It represents all types and severities of disability.

The objective of this study is to describe the level of leisure physical activity of people who are members or users of APF France handicap and their barriers to physical activity.

DETAILED DESCRIPTION:
This is a national transversal study aiming at studying the level of leisure physical activity among people with disabilities, members or users of APF France handicap.

The study is based on a survey by questionnaire to the APF France handicap community. The survey is distributed between April and June 2023 through a public communication campaign (emails, posters, website, social networks, etc.). Data on leisure physical activity, barriers to physical activity and quality of life will be collected.

The questionnaire has been translated in simplified French to facilitate its understanding.

This is a survey that collects data anonymously and follows the MR004 methodology.

ELIGIBILITY:
Inclusion Criteria:

* Members or users of APF France handicap
* People with disability
* Agreeing to participate in the survey

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members or users of APF France handicap.
Sampling Method: Non-Probability Sample
Enrollment: 769 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | Baseline
  Physical Activity Scale for Individuals with Physical Disabilities (PASIPD) Questionnaire - Leisure Time Activity Section

SECONDARY OUTCOMES:
Barriers of physical activity | Baseline
  Barriers to Physical Activity Questionnaire for People with Mobility Impairments. Modified version by a group of experts, including representatives of the APF France handicap. Version not detailing the importance of each barrier.
Quality of life | Baseline
  EuroQol EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Carpentier, MD-MSc, Study Chair — ISPC Synergies; François Genêt, MD-PhD, Principal Investigator — ISPC Synergies
Locations (1):
- ISPC Syngergies, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided